CLINICAL TRIAL: NCT05246007
Title: Effect of Nocturnal Low-dose Dexmedetomidine Infusion on Sleep Quality in Older Patients Undergoing Knee or Hip Replacement Surgery: A Multicenter Randomized Controlled Trial
Brief Title: Nocturnal Low-dose Dexmedetomidine Infusion and Perioperative Sleep Quality
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We changed the protocol and registered for another trial.
Sponsor: Peking University First Hospital (Other)
Collaborators: Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2021-639
Record Dates: First submitted 2022-02-08; First posted 2022-02-18 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Old Age; Knee Replacement Surgery; Hip Replacement Surgery; Dexmedetomidine; Sleep Quality
Keywords: Old Age; Knee replacement surgery; Hip replacement surgery; Dexmedetomidine; Sleep quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Experimental): Dexmedetomidine will be infused at a rate of 0.02 ml/kg/h (0.025 μg/kg/h) during the night before surgery, the night of surgery, and the first 2 nights after surgery (from 9:00 pm-6:00 am).
  Interventions: Drug: Dexmedetomidine
- Placebo group (Placebo Comparator): Placebo (normal saline) will be infused at a rate of 0.02 ml/kg/h during the night before surgery, the night of surgery, and the first 2 nights after surgery (from 9:00 pm-6:00 am).
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine will be infused at a rate of 0.02 ml/kg/h (0.025 μg/kg/h) during the night before surgery, the night of surgery, and the first 2 nights after surgery (from 9:00 pm-6:00 am).
  Other Names: Dexmedetomidine for infusion
  Arms: Dexmedetomidine group
Drug: Normal Saline — Placebo (normal saline) will be infused at a rate of 0.02 ml/kg/h during the night before surgery, the night of surgery, and the first 2 nights after surgery (from 9:00 pm-6:00 am).
  Other Names: Normal Saline for infusion
  Arms: Placebo group

SUMMARY:
Sleep disturbances are prevalent in older patients with osteoarthrosis or fracture scheduled for knee or hip replacement surgery. The occurrence of sleep disturbances is associated with worse outcomes including increased risk of delirium and cardiac events, and worsened functional recovery. Dexmedetomidine is a highly selective α2-adrenergic agonist with sedative, anxiolytic, and analgesic properties. It exerts sedative effects via activating the endogenous sleep pathways and produces a state like non-rapid eye movement sleep, which is different from opioid- and benzodiazepine-induced sedation. Night-time infusion of low-dose dexmedetomidine may improve sleep quality. However, evidence in this aspect is limited.

DETAILED DESCRIPTION:
Sleep is a naturally recurring state characterized by lowered consciousness, reduced sensory and voluntary activity, and inhibited interaction with surroundings. Normal sleep has a particular structure and significant circadian rhythms; and is vital for both physical and mental health. Evidence shows that the restorative effect of sleep may be a consequence of the enhanced removal of potentially neurotoxic waste products like β-amyloid or tau protein via the glymphatic pathway in the neurological system.

Sleep disturbances frequently occur in elderly patients with chronic pain and complicated comorbidity. A meta-analysis shows that in adults, total sleep time, sleep efficiency, percentage of slow-wave sleep, and percentage of rapid eye movement (REM) sleep significantly decrease, while sleep latency, percentage of stage 1 non-REM sleep, percentage of stage 2 non-REM sleep, and wake after sleep onset significantly increase with ageing. Coexisting disease such as asthma and obstructive sleep apnea are also associated with poorer sleep quality, as manifested by increased stage 1 and 2 non-REM sleep, and decreased REM sleep. Furthermore, pain and sleep disturbances are closely correlated, and sleep disturbances frequently accompany pain from osteoarthritis (OA) or fracture in elderly patients who are scheduled for knee or hip arthroplasty.

Sleep disturbances are common after major surgery owing to preoperative comorbidity, residual anesthetic effects, surgical trauma, postoperative pain, use of analgesics, and hospital environment. Patients may report shortened total sleep time, increased number of arousals/awakenings, lowered subjective sleep quality, and sometimes nightmares. Polysomnographic monitoring reveals sleep deprivation, sleep fragmentation, altered sleep architecture (increased light sleep, decreased or disappeared deep and rapid eye movement sleep), and disordered circadian rhythm. Considering the importance of normal sleep for human health, it is not surprising that sleep disturbances may produce harmful effects on patients' recovery. Indeed, emerging evidence suggests that sleep disturbances are associated with increased sensitivity to pain, higher inflammation, more delirium, more cardiovascular events, and prolonged hospital stay.

Dexmedetomidine, an α2 adrenoceptor agonist with both sedative and analgesic properties, has increasingly been used. Unlike other sedative agents, dexmedetomidine exerts its sedative effects through an endogenous sleep-promoting pathway and preserves sleep architecture to some degree. In a recent study of mechanically ventilated ICU patients, nighttime infusion of a sedative dose of dexmedetomidine (median infusion rate 0.6 μg/kg/h [interquartile range, 0.4 to 0.7]) helped preserve the circadian of sleep and improved the sleep architecture by increasing sleep efficiency and stage 2 non-REM sleep. In our previous study of non-mechanically ventilated ICU patients, nighttime infusion of low-dose of dexmedetomidine (0.1 μg/kg/h) improved the sleep architecture by increasing sleep efficiency and stage 2 non-REM sleep. Our subsequent large randomized controlled trial showed that low-dose night-time infusion of dexmedetomidine improved sleep and decreased the incidence of delirium; furthermore, it improved 2-year survival and 3-year quality of life after surgery.

We suppose that, for older patients with osteoarthrosis or fracture who are scheduled for knee or hip replacement surgery, nighttime infusion of low-dose dexmedetomidine starting from the preoperative night and continuing in the postoperative period may improve sleep quality and postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years and <90 years;
* Scheduled to undergo unilateral knee or hip arthroplasty under spinal or combined spinal-epidural anesthesia.

Exclusion Criteria:

* Refuse to participate;
* Hypnotic therapy for sleep disorders within 3 months;
* Presence of contraindications to intrathecal anesthesia;
* Preoperative history of schizophrenia, epilepsy, Parkinson's disease, myasthenia gravis, or delirium;
* Diagnosed as obstructive sleep apnea, or at high risk of moderate to severe obstructive sleep apnea according to the STOP-Bang questionnaire;
* Inability to communicate in the preoperative period because of coma, profound dementia, or language barrier;
* Sick sinus syndrome, severe sinus bradycardia (heart rate <50 beats/min), or atrioventricular block above grade II without pacemaker implanted;
* Severe hepatic dysfunction (Childe Pugh class C); renal dysfunction (required preoperative dialysis), or expected survival ≤24 hours;
* Receiving treatment with dexmedetomidine or clonidine;
* Allergy to dexmedetomidine.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Subjective sleep quality (overall RCSQ score) during the night of surgery. | During the night of surgery.
  Subjective sleep quality will be assessed in the morning (between 8:00 am to 10:00 am) using the Richards-Campbell Sleep Questionnaire (RCSQ). The RCSQ is a self-reported measure that evaluated perception of nighttime sleep in five items, including sleep depth, sleep latency, number of awakenings, returning to sleep, and overall sleep quality. Each item was assessed with a 100-millimeter visual analog scale (VAS; score ranges from 0 to 100, with higher scores representing better sleep). The mean score of the five items represents the overall RCSQ score. The RCSQ also included a sixth item, not included in the overall score, that evaluated perceived nighttime noise (score ranges from 0 to 100, where 0="very noisy" and 100="very quiet").

SECONDARY OUTCOMES:
Subjective sleep quality (overall RCSQ score) during the perioperative period. | From the night before surgery until the fifth night after surgery.
  Subjective sleep quality will be assessed daily in the morning (between 8:00 am to 10:00 am) using the Richards-Campbell Sleep Questionnaire (RCSQ).
Total sleep time per night during the perioperative period. | From the night before surgery until the fifth night after surgery.
  Objective sleep quality will be monitored with an actigraphy from 6:00 pm to 8:00 am from the night before surgery until the fifth night after surgery. Total sleep time is defined as the sum in time scored as asleep.
Sleep efficiency per night during the perioperative period. | From the night before surgery until the fifth night after surgery.
  Objective sleep quality will be monitored with an actigraphy from 6:00 pm to 8:00 am from the night before surgery until the fifth night after surgery. Sleep efficiency is defined as 100*total sleep time/time in bed.
Sleep onset latency per night during the perioperative period. | From the night before surgery until the fifth night after surgery.
  Objective sleep quality will be monitored with an actigraphy from 6:00 pm to 8:00 am from the night before surgery until the fifth night after surgery. Sleep onset latency is defined as time difference between time to bed and sleep start.
Wake after sleep onset per night during the perioperative period. | From the night before surgery until the fifth night after surgery.
  Objective sleep quality will be monitored with an actigraphy from 6:00 pm to 8:00 am from the night before surgery until the fifth night after surgery. Wake after sleep onset is defined as the total time scored as awake between sleep start and sleep end.
Intensity of pain during the first 3 postoperative days. | Up to 3 days after surgery.
  Intensity of pain will be assessed at 6, 12, 24, 48, and 72 hours after surgery with the Numeric Rating Scale (an 11-point scale where 0 indicates no pain and 10 the worst pain)
The incidence of delirium within 5 days after surgery. | Up to 5 days after surgery.
  Delirium is assessed twice daily (8:00-10:00 am and 6:00-8:00 pm) with the 3-minute diagnostic interview for Confusion Assessment Method-defined delirium (3D-CAM).
The joint range of motion after surgery. | Up to 5 days after surgery.
  Range of motion is assessed between 8:00 am to 10:00 am at 1, 3, and 5 days after surgery.
Length of stay in hospital after surgery. | Up to 30 days after surgery.
  Length of stay in hospital after surgery.
Incidence of non-delirium complications within 30 days. | Up to 30 days after surgery.
  Non-delirium complications are defined as newly occurred medical events other than delirium that are deemed harmful and required therapeutic intervention, i.e., grade II or higher on the Clavien-Dindo classification.
Subjective sleep quality (Pittsburgh Sleep Quality Index) at 30 days after surgery. | On the 30th day after surgery.
  Subjective sleep quality at 30 days after surgery will be assessed with the Pittsburgh Sleep Quality Index. This is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score.
Cognitive function at 3 months after surgery. | At the end of the 3rd month after surgery.
  Cognitive function is assessed with the modified Telephone Interview for Cognitive Status.
Quality of life at 3 months after surgery. | At the end of the 3rd month after surgery.
  Quality of life is assessed with short form 36 questionnaire.
3-year overall survival. | Up to 3 years after surgery.
  Overall survival is defined as the time interval from surgery to all-cause death.
3-year event-free survival. | Up to 3 years after surgery.
  Event-free survival is defined as the time interval from surgery to the earliest date of new serious disease (require hospitalization) or all-cause death.
Cognitive function within 3 years after surgery. | Up to 3 years after surgery.
  Cognitive function will be assessed at the end of each year after surgery, with the modified Telephone Interview for Cognitive Status.
Quality of life every year within 3 years after surgery. | Up to 3 years after surgery.
  Quality of life will be assessed at the end of each year after surgery, with short form 36 questionnaire.

OTHER OUTCOMES:
Cerebrospinal fluid proteomics examination (selected patients). | During anesthesia.
  Cerebrospinal fluid (1 ml) will be collected during spinal anesthesia. Deep proteome analysis will be performed to detect protein biomarkers including amyloid-beta, total tau, and phosphorylated tau.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (2):
- China (2):
  - Beijing Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel JM. Sleep viewed as a state of adaptive inactivity. Nat Rev Neurosci. 2009 Oct;10(10):747-53. doi: 10.1038/nrn2697. Epub 2009 Aug 5. PMID 19654581
- [Background] Xie L, Kang H, Xu Q, Chen MJ, Liao Y, Thiyagarajan M, O'Donnell J, Christensen DJ, Nicholson C, Iliff JJ, Takano T, Deane R, Nedergaard M. Sleep drives metabolite clearance from the adult brain. Science. 2013 Oct 18;342(6156):373-7. doi: 10.1126/science.1241224. PMID 24136970
- [Background] Onen SH, Onen F, Courpron P, Dubray C. How pain and analgesics disturb sleep. Clin J Pain. 2005 Sep-Oct;21(5):422-31. doi: 10.1097/01.ajp.0000129757.31856.f7. PMID 16093748
- [Background] Lintzeris N, Moodley R, Campbell G, Larance B, Bruno R, Nielsen S, Degenhardt L. Sleep Quality Among People Living With Chronic Noncancer Pain: Findings From the Pain and Opioids IN Treatment (POINT) Cohort. Clin J Pain. 2016 May;32(5):380-7. doi: 10.1097/AJP.0000000000000282. PMID 26218004
- [Background] Er MS, Altinel EC, Altinel L, Erten RA, Eroglu M. An assessment of sleep quality in patients undergoing total knee arthroplasty before and after surgery. Acta Orthop Traumatol Turc. 2014;48(1):50-4. doi: 10.3944/AOTT.2014.3163. PMID 24643100
- [Background] Sasaki E, Tsuda E, Yamamoto Y, Maeda S, Inoue R, Chiba D, Okubo N, Takahashi I, Nakaji S, Ishibashi Y. Nocturnal knee pain increases with the severity of knee osteoarthritis, disturbing patient sleep quality. Arthritis Care Res (Hoboken). 2014 Jul;66(7):1027-32. doi: 10.1002/acr.22258. PMID 24470323
- [Background] Fatah RMN, Abdulrahman BB. A sleep disturbance after total knee arthroplasty. J Family Med Prim Care. 2020 Jan 28;9(1):119-124. doi: 10.4103/jfmpc.jfmpc_595_19. eCollection 2020 Jan. PMID 32110576
- [Background] Alexopoulou C, Kondili E, Diamantaki E, Psarologakis C, Kokkini S, Bolaki M, Georgopoulos D. Effects of dexmedetomidine on sleep quality in critically ill patients: a pilot study. Anesthesiology. 2014 Oct;121(4):801-7. doi: 10.1097/ALN.0000000000000361. PMID 24988068
- [Background] Wu XH, Cui F, Zhang C, Meng ZT, Wang DX, Ma J, Wang GF, Zhu SN, Ma D. Low-dose Dexmedetomidine Improves Sleep Quality Pattern in Elderly Patients after Noncardiac Surgery in the Intensive Care Unit: A Pilot Randomized Controlled Trial. Anesthesiology. 2016 Nov;125(5):979-991. doi: 10.1097/ALN.0000000000001325. PMID 27571256
- [Background] Su X, Meng ZT, Wu XH, Cui F, Li HL, Wang DX, Zhu X, Zhu SN, Maze M, Ma D. Dexmedetomidine for prevention of delirium in elderly patients after non-cardiac surgery: a randomised, double-blind, placebo-controlled trial. Lancet. 2016 Oct 15;388(10054):1893-1902. doi: 10.1016/S0140-6736(16)30580-3. Epub 2016 Aug 16. PMID 27542303
- [Background] Zhang DF, Su X, Meng ZT, Li HL, Wang DX, Xue-Ying Li, Maze M, Ma D. Impact of Dexmedetomidine on Long-term Outcomes After Noncardiac Surgery in Elderly: 3-Year Follow-up of a Randomized Controlled Trial. Ann Surg. 2019 Aug;270(2):356-363. doi: 10.1097/SLA.0000000000002801. PMID 29742525
- [Background] Li HJ, Li CJ, Wei XN, Hu J, Mu DL, Wang DX. Dexmedetomidine in combination with morphine improves postoperative analgesia and sleep quality in elderly patients after open abdominal surgery: A pilot randomized control trial. PLoS One. 2018 Aug 14;13(8):e0202008. doi: 10.1371/journal.pone.0202008. eCollection 2018. PMID 30106963